CLINICAL TRIAL: NCT06311370
Title: Acceptability, Feasibility, and Development of an AI Driven, Multi-sensor, Non-invasive Digital Mental Health Platform in Children With ADHD and Emotional Symptoms
Status: Completed | Type: Observational
Sponsor: MaxisHealth (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-0100
Record Dates: First submitted 2024-02-20; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: ADHD; Autism
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Autistic Disorder | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children age 4 to 7: Children age 4-7 in therapeutic school, diagnosed with ADHD, Autism monitored with raters and the sensor watch.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observed by trained staff and wearing a sensor watch

SUMMARY:
This is an observational study collecting data using a wearable to measure the biometric features in youth with Attention deficit hyperactivity disorder(ADHD) and Autism.

DETAILED DESCRIPTION:
Participants in therapeutic school for disruptive behavior with Attention deficit hyperactivity disorder( ADHD), Autism with age 4-7 year old. Participant will wear watch during their school days for 5 days in presence of investigator and raters taking behavioral observation. The data collected from the raters and wearable will be analyzed to correlate emotional dysregulation.

ELIGIBILITY:
Inclusion Criteria:

* Children in the therapeutic school, diagnosed with ADHD

Exclusion Criteria:

* Unable to tolerate wearing the watch

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with ADHD attending the therapeutic school.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Emotion dysregulation | 20 hours upto 4 weeks
  Number of tantrums

CONTACTS AND LOCATIONS:
Locations (1):
- The League School, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No